CLINICAL TRIAL: NCT03071731
Title: Glittre Activities of Daily Life-test: Responsiveness to Acute Bronchodilation in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Glittre ADL-test: Responsiveness to Acute Bronchodilation in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: Glittre
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Didier Saey, Researcher-Associate Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2017-2739
Record Dates: First submitted 2017-02-16; First posted 2017-03-07 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Glittre; COPD; sit-to-stand; responsiveness; bronchodilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchodilator Agents; Ipratropium; Albuterol

STUDY DESIGN:
Intervention Model Description: Participants receive one intervention (bronchodilation before performing a functional test) during the initial phase of the study and during the second phase of the study are evaluated in parallel after receiving a placebo or vice versa (random order)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization to decide on which visit the participant will receive the placebo will be generated by a software and managed by the main investigator. Bronchodilators and the placebo will be put in an aerosol of same shape and color so the participants and outcomes assessor won't be able to tell which one is which.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchodilators (Experimental): Nebulization of ipratropium bromide/salbutamol sulfate (500 µg/2.5 mg) before the administration of the Glittre ADL-test
  Interventions: Drug: Bronchodilators; Drug: Placebos
- Placebo (Placebo Comparator): Nebulization of a placebo before the administration of the Glittre ADL-test
  Interventions: Drug: Bronchodilators; Drug: Placebos

INTERVENTIONS:
Drug: Bronchodilators — Administration of a nebulized combination of bronchodilators before the administration of a functional test.
  Other Names: ipratropium bromide; salbutamol sulfate
Drug: Placebos — Administration of a nebulized placebo before the administration of a functional test
  Other Names: nebulized placebo

SUMMARY:
This project is aimed to assess the responsiveness of the Glittre ADL-test and the 1-Minute Sit-to-Stand test (1-Minute STST) to acute bronchodilation in patients with COPD. We also aim to investigate the physiological and perceptual response to bronchodilation of the Glittre ADL-test and the 1-minute STST. The specific objectives are 1)To measure the changes in time for completion of the Glittre ADL-test and the number of standing up during the 1-minute STST induced by a single dose of nebulized ipratropium bromide/salbutamol sulfate against those induced by a placebo in patients with moderate to severe COPD and 2)To compare in patients with moderate to severe COPD the CR (minute ventilation (VE), oxygen uptake (VO2), carbon dioxide production (VCO2) and heart rate) and symptomatic (dyspnea and leg fatigue perception) responses during the Glittre ADL-test and the 1-Minute STST following a single dose of ipratropium bromide/salbutamol sulfate or placebo. We suppose among others that the Glittre test completion time will be lesser, that the number of repetitions in the 1-Minute STST will be higher and symptoms intensity will be lesser among patients with COPD receiving bronchodilators.

DETAILED DESCRIPTION:
METHODOLOGY: Study design and setting: It will be a randomized double-blind trial during which 34 patients with moderate to severe COPD will complete 2 Glittre ADL-tests 15 minutes following nebulization of a placebo or of ipratropium bromide/salbutamol sulfate combination. Patients receiving bronchodilators before the beginning of the study will be asked to withdraw from their medication 8h in the case of short-acting bronchodilators and/or 72 h in the case of long-acting bronchodilators before visits. Those treated with tiotropium will have a 4-week washout period during which this therapy will be replaced by ipratropium bromide. The study will require 3 visits to the research center of Institut Universitaire de Cardiologie et de Pneumologie de Québec-Université Laval (IUCPQ). The 1st visit will be devoted to verify the eligibility to the study, obtain informed consent, and measure baseline characteristic including anthropometric measurements, pulmonary, and lower limb muscle function, as well maximal exercise capacity and participation in activities of daily life. In addition, participants will be familiarized with the Glittre test. During the following visits, subjects will complete two Glittre tests (1/visit) preceded by administration of nebulized placebo or ipratropium bromide/salbutamol sulfate (500 mg/2.5 mg) administrated in a randomized and double-blind fashion. Study visits will be separated by >72 h and <7 days. Subjects will be scheduled to attend at the same time of day throughout the study. Ethics approval will be obtained before starting the project and all subjects will provide written informed consent prior to testing. Procedure and measurements: Anthropometric measurements: Weight and height will be measured on a standing scale. Pulmonary function: Complete pulmonary function tests including spirometry, lung volumes and diffusing capacity for carbon monoxide will be obtained according to standardized technique and expressed as a percent of predicted9. In addition, during visit 2 and 3, a spirometry (FEV1 and FVC) will be obtained before and after bronchodilation to determine bronchodilator-induced change in FEV1 and baseline respiratory condition before functional tests. Muscle function: Quadriceps muscle function (force, endurance and fatigue) will be quantified during a knee extension test. The test will consist of one set of 30 repetitions at an angular velocity of 90°/s. Amplitude and angular velocity will be controlled using a dynamometric isokinetic system (Biodex, system pro 4, Biodex Medical System, Shirley, NY, USA). Maximal exercise capacity: Maximal exercise capacity will be assessed using a symptom-limited incremental cycling test. Subjects will be seating on an electrically braked ergocycle (Quinton Corival 400; A-H Robins, Seattle, WA) and connected to a portable a gas analysis system (Oxycon Mobile, Viasys Healthcare, Jaeger, Germany). After 5 minutes of rest, a progressive stepwise exercise test will be performed up to the individual maximal capacity. Each exercise step lasts 1 minute and increments of 10 watts will be applied. Minute ventilation (VE), oxygen uptake (VO2), and CO2 excretion (VCO2) respiratory exchange ratio (RER), respiratory rate (RR) inspiratory capacity (IC) and heart rate (HR) will be measured at rest and during exercise on a breath-by-breath basis. In addition, pulsed oxygen saturation (SpO2) will be measured at rest, continuously during the tests, and at end-exercise by pulse oximetry (OSM2 Hemoximeter; Radiometer,Copenhagen, Denmark). Dyspnea and leg fatigue perception will be measured by a modified Borg scale at rest, each 2 minutes and at the end of exercise. Participation in activities of daily life: Participation in activities of daily life will be measured with an accelerometer-based activity monitor (DynaPort Minimod, McRoberts BV, The Hague, The Netherlands). Patients will be instructed to wear the monitor on the waist for 7 consecutive days. They will also fill a diary of activities through the week they are wearing the physical activity monitor. Self-efficacy: Patients' perceived walking and climbing stairs confidence (on flat ground, with and without handrail) will be assessed with the 10-item self-report modified Gait Efficacy Scale. Functional tests: The Glittre ADL tests will be completed according to the original procedure described by Skumlien5. Briefly, patient carrying a weighted backpack (2.5 kg for women, 5.0 kg for men) will be instructed to stand up and walk along a flat 10-m long course. In the middle of the course, there will be a 2-step staircase (each step 17 cm high×27 cm deep) to get across. After completing the second 5 m, the subject will be facing a shelf containing 3 objects, each weighing 1 kg, positioned on the top shelf (shoulder height). Participants will then move objects, 1 by 1, to the bottom shelf (waist height) and then to the floor. Once completed, participants will then have to return the objects, always 1 by 1, to the bottom shelf and finally to the top shelf again. Participants will then walk back along the circuit, climbing and descending the stairs, until reaching the starting point (chair); sitting down and immediately beginning the next lap. Patients will be instructed to complete 5 laps on this circuit as quickly as possible. The 1-minute STST will be completed according to the procedure described by Ozalevli and al. Patients will be instructed to fully stand up from a chair, arms across the chest, sit back down and repeat as often as possible during one minute. Physiological measures as well as dyspnea and leg fatigue perception will be acquired with the same methodology used for the maximal exercise capacity. The order of functional tests will be randomized for each patient. Patients will also fill the Multidimensional Dyspnea Profile questionnaire. Global rating of change: Patients' perception of change in their performance, dyspnea and leg fatigue induced by the functional tests will be ascertain with a 7-point Likert Scale ranging from -3 (large deterioration) to +3 (large improvement) immediately after each functional test. No feedback from the evaluator will be given to patients before patients' own rating.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe COPD based on the GOLD spirometric classification
* able to provide written informed consent
* able to follow verbal directions for testing.

Exclusion Criteria:

* diagnosed with cardiovascular, neurological or, neuromuscular conditions that could affect ability to perform the tests (e.g. stroke, knee osteoarthritis);
* currently participating in a structured exercise or pulmonary rehabilitation program or been involved in pulmonary rehabilitation in the past 6 months;
* experienced a COPD exacerbation in the past 6 weeks
* receiving a daily dose > 10mg of oral Prednisone within the past 3 months
* unable to walk 4 metres without use of a gait aid (e.g. walker, cane)
* receiving oxygen supply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Glittre ADL-test time completion | Between 2 and 12 minutes for each test; up to three days between the two tests
  Time to complete 5 laps as fast as possible

SECONDARY OUTCOMES:
Perceptual variables | Up to three days between the two administrations
  Dyspnea and fatigue in the legs at the end of the Glittre ADL-test
Perceptual variables | Up to three days between the two administrations
  Dyspnea and fatigue in the legs at the end of the 1-minute STST
Breathing discomfort | Up to three days between the two administrations
  Overall subjective experience of breathing discomfort after the Glittre ADL-test assessed with the Multidimensional Dyspnea Profile questionnaire
Breathing discomfort | Up to three days between the two administrations
  Overall subjective experience of breathing discomfort after the 1-minute STST assessed with the Multidimensional Dyspnea Profile questionnaire
Accelerometry-subduration | Up to three days between the two administrations
  Subduration (in seconds) in the Glittre ADL-test for each component, in each lap
Accelerometry-steps | Up to three days between the two administrations
  Number of steps in the Glittre ADL-test for each walking section, in each lap
Accelerometry | Up to three days between the two administrations
  Vertical and horizontal acceleration and deceleration (m/s) in the Glittre ADL-test for each component, in each lap
Accelerometry | Up to three days between the two administrations
  Vertical and horizontal acceleration and deceleration (m/s) in the 1-minute STST for each repetition.
Hyperinflation | Between 2 and 12 minutes for the IC measures at the beginning and at the end of the Glittre test, and up to 3 days before the 2nd assessment
  Change of IC between the beginning and end of the Glittre ADL-test completed after the administration of the placebo compared with the change of IC between the beginning and end of the Glittre test after the administration of the combination of bronchodilators
Hyperinflation | In a 5-minute time frame for the IC measures at the beginning and at the end of the 1-minute STST, and up to 3 days before the 2nd assessment
  Change of IC between the beginning and end of the 1-minute STST completed after the administration of the placebo compared with the change of IC between the beginning and end of the 1-minute STST after the administration of the combination of bronchodilators
Physiological variable-ventilation | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first Glittre ADL-test, and up to 13 days between the test on the bike and the 2nd Glittre ADL-test
  Minute ventilation (VE; L/min) during the two Glittre ADL-test compared to the VE during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variable-ventilation | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first 1-minute STST, and up to 13 days between the test on the bike and the 2nd 1-minute STST
  Minute ventilation (VE; L/min) during the two 1-minute STST compared to the VE during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variable-ratio exchange rate | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first Glittre ADL-test, and up to 13 days between the test on the bike and the 2nd Glittre ADL-test
  Ratio exchange rate (RER) the two Glittre ADL-tests compared to RER during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variable-ratio exchange rate | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first 1-minute STST, and up to 13 days between the test on the bike and the 2nd 1-minute STST
  Ratio exchange rate (RER) the two 1-minute STST compared to RER during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variables-VO2 and VCO2 | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first Glittre ADL-test, and up to 13 days between the test on the bike and the 2nd Glittre ADL-test
  VO2 and VCO2 during the two Glittre ADL-tests compared to those during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variables-VO2 and VCO2 | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first 1-minute STST, and up to 13 days between the test on the bike and the 2nd 1-minute STST
  VO2 and VCO2 during the two 1-minute STST compared to those during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variable-HR | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first Glittre ADL-test, and up to 13 days between the test on the bike and the 2nd Glittre ADL-test
  Peak Heart rate (HR; beats/minute) during the two Glittre ADL-test compared to peak heart rate during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variable-HR | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first 1-minute STST, and up to 13 days between the test on the bike and the 2nd 1-minute STST
  Peak Heart rate (HR; beats/minute) during the two 1-minute STST compared to peak heart rate during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variable-RR | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first Glittre ADL-test, and up to 13 days between the test on the bike and the 2nd Glittre ADL-test
  Peak respiratory rate (breaths/min) during the two Glittre ADL-test compared to peak heart rate during an incremental cardiopulmonary maximal exercise test on bike.
Physiological variable-RR | Up to 10 days between the cardiopulmonary maximal exercise test on the bike and the first 1-minute STST, and up to 13 days between the test on the bike and the 2nd 1-minute STST
  Peak respiratory rate (breaths/min) during the two 1-minute STST compared to peak heart rate during an incremental cardiopulmonary maximal exercise test on bike.
Number of repetitions 1-Minute STST | About 2-3 minutes for test administration including instructions and demonstration; up to 3 days between both administration
  Number of full stand-up repetitions in the 1-Minute STST in both conditions (following the administration of the placebo and the bronchodilators)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Saey, Ph.D., Principal Investigator — Centre de recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Québec
Locations (1):
- Centre de recherche-Institut Universitaire de Cardiologie et Pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participant data sets on characterization (muscle and pulmonary function, cardiopulmonary exercise testing) and medical history collected during the recruitment interview will be made available to other researchers after the end of the study, upon request. Data will be obtained through electronical denominalized files.

REFERENCES:
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Velloso M, Stella SG, Cendon S, Silva AC, Jardim JR. Metabolic and ventilatory parameters of four activities of daily living accomplished with arms in COPD patients. Chest. 2003 Apr;123(4):1047-53. doi: 10.1378/chest.123.4.1047. PMID 12684292
- [Background] Annegarn J, Meijer K, Passos VL, Stute K, Wiechert J, Savelberg HH, Schols AM, Wouters EF, Spruit MA; Ciro+ Rehabilitation Network. Problematic activities of daily life are weakly associated with clinical characteristics in COPD. J Am Med Dir Assoc. 2012 Mar;13(3):284-90. doi: 10.1016/j.jamda.2011.01.002. Epub 2011 Feb 17. PMID 21450242
- [Background] Skumlien S, Hagelund T, Bjortuft O, Ryg MS. A field test of functional status as performance of activities of daily living in COPD patients. Respir Med. 2006 Feb;100(2):316-23. doi: 10.1016/j.rmed.2005.04.022. Epub 2005 Jun 6. PMID 15941658
- [Background] Karloh M, Karsten M, Pissaia FV, de Araujo CL, Mayer AF. Physiological responses to the Glittre-ADL test in patients with chronic obstructive pulmonary disease. J Rehabil Med. 2014 Jan;46(1):88-94. doi: 10.2340/16501977-1217. PMID 24104462
- [Background] Correa KS, Karloh M, Martins LQ, dos Santos K, Mayer AF. Can the Glittre ADL test differentiate the functional capacity of COPD patients from that of healthy subjects? Rev Bras Fisioter. 2011 Nov-Dec;15(6):467-73. doi: 10.1590/s1413-35552011005000034. Epub 2011 Nov 21. English, Portuguese. PMID 22094546
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] Ribeiro F, Lepine PA, Garceau-Bolduc C, Coats V, Allard E, Maltais F, Saey D. Test-retest reliability of lower limb isokinetic endurance in COPD: A comparison of angular velocities. Int J Chron Obstruct Pulmon Dis. 2015 Jun 18;10:1163-72. doi: 10.2147/COPD.S81806. eCollection 2015. PMID 26124656
- [Background] Langer D, Gosselink R, Sena R, Burtin C, Decramer M, Troosters T. Validation of two activity monitors in patients with COPD. Thorax. 2009 Jul;64(7):641-2. doi: 10.1136/thx.2008.112102. No abstract available. PMID 19561287
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893